CLINICAL TRIAL: NCT02856633
Title: Preliminary Testing of the Vitaliti CVSM Wearable, Vitaliti Spirotoscope, and Vitaliti IVD Station
Status: Completed | Type: Observational
Sponsor: Cloud DX Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: STP-VIT-001
Record Dates: First submitted 2016-07-29; First posted 2016-08-05 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Urinary Tract Infection; Diabetes Mellitus; Atrial Fibrillation; OSA; COPD; Pneumonia; Acute Otitis Media; Leukocytosis; Iron Deficient Anemia; Hypertension; Healthy Volunteers
MeSH Terms: conditions — Urinary Tract Infections; Diabetes Mellitus; Atrial Fibrillation; Pulmonary Disease, Chronic Obstructive; Pneumonia; Otitis Media; Leukocytosis; Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vitaliti System
  Interventions: Device: Vitaliti

INTERVENTIONS:
Device: Vitaliti

SUMMARY:
The study objective is to satisfy the testing requirements for the Qualcomm Tricorder XPRIZE Competition. This requires an oversight model using the Vitaliti CVSM Wearable, Vitaliti Spirotoscope, and Vitaliti IVD Station to continuously monitor the patient's five core vital signs and to detect the health conditions required by the competition.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years of age.
* English speaking
* Established diagnosis of one of the thirteen required conditions with evidence in Medical Record.

Exclusion Criteria:

* Lack of patient consent
* Has pacemaker or internal medical device
* Pregnancy
* Concurrent enrollment into a clinical trial that may affect subject treatment
* Age less than 18 or over 65
* Physical disabilities affecting vision (eyeglasses or contact lenses will be allowed), manual manipulation, or use of a computer or mobile device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult subjects with urinary tract infection, diabetes mellitus, atrial fibrillation, sleep apnea, COPD, pneumonia, acute otitis media, leukocytosis, anemia, or hypertension will be recruited to participate in this observational study from Oakville-Trafalgar Memorial Hospital.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-02-19 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Successful diagnosis of patient's condition by Vitaliti software as compared to patient's Medical Record | 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Sonny Kohli, MD, Principal Investigator — Oakville Trafalgar Memorial Hospital
Locations (1):
- Oakville Trafalgar Memorial Hospital, Oakville, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No